CLINICAL TRIAL: NCT03031483
Title: A Phase II Trial Addressing Feasibility and Activity of Clarithromycin + Lenalidomide Combination: a Full Oral Treatment for Patients With Relapsed/Refractory Extranodal Marginal Zone Lymphoma
Brief Title: Clarithromycin + Lenalidomide Combination: a Full Oral Treatment for Patients With Relapsed/Refractory Extranodal Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG40
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Mucosa Associated Lymphoid Tissue (MALT) Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Clarithromycin; Lenalidomide

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: clarithromycin and lenalidomide (Experimental): CLARITHROMYCIN: daily orally administration in cycles of 28 days; 500mg film-coated tablets LENALIDOMIDE: every cycle of treatment lasts 28 days; daily orally administration is of 21 consecutive days with a week of rest. 20mg capsule hard. The maximum treatment duration is 12 months.
  Interventions: Drug: clarithromycin and lenalidomide

INTERVENTIONS:
Drug: clarithromycin and lenalidomide — Each treatment course will consist of:
  Oral Lenalidomide (Revlimid) once daily for 21 days at a dose 20 mg; in case of drug-related adverse events the dose can be reduced to 15 and 10 mg/day; Oral Clarithromycin 500 mg twice daily for 28 days. Courses will be repeated every 28 days. After the first 3 courses patients with stable disease or better response will be given another three courses. Patients with complete remission or disease progression after 6 courses will be taken off study, while patients with partial response or stable disease will receive 3 further courses of treatment. Again, patients with complete response or disease progression will stop therapy, while patients with partial response/stable disease will receive 3 further courses up to a maximum of 12 courses in total.

SUMMARY:
Patients with lymphoid tissue lymphoma mucosa-associated (MALT) for which the standard treatments with radiotherapy, chemotherapy and / or immunotherapy show lack of efficacy

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified diagnosis of MALT lymphoma arising at any extranodal site
* Disease refractory to or in first or greater relapse after prior radiotherapy and/ or chemotherapy and/or immunotherapy
* Measurable or non-measurable lesions where the response is nevertheless evaluable by non-imaging means (e.g., gastric or bone marrow infiltrations)
* Ann Arbor Stage I-IV
* ECOG performance status of 0, 1 or 2
* Age ≥ 18 years
* Life expectancy of at least 3 months
* Adequate haematological status: ANC (absolute neutrophil count [segmented + bands]) ≥1.0 x 109/L, platelet count ≥ 75 x 109/L , haemoglobin ≥8 g/dL.
* Adequate cardiac, renal and liver function tests (LVEF > 40%, serum creatinine < 2.5 mg/dl, ALAT or ASAT < 2.5 x upper limit of normal range, alkaline phosphatase < 2.5 x upper limit of normal range, serum bilirubin < 2.0 mg/dl)
* Patient must be willing and able to comply with the protocol for the entire study duration
* Female patients of childbearing potential must agree to use, and be able to comply with, effective contraception and agree to have medically supervised pregnancy tests prior to starting the study treatment and during therapy
* Male patients must agree to always use a condom during any sexual contact with females of reproductive potential and agree to not donate sperm while taking lenalidomide
* Patient must agree to abstain from donating blood while taking study drug therapy
* Patient must agree not to share study medication with another person and to return all unused study drug to the investigator
* Patient must be willing and able to comply with the protocol
* Patient must be capable of understanding

Exclusion Criteria:

* Lymphoma histology other than MALT lymphoma or MALT lymphoma with a diffuse large cell lymphoma ("high grade lymphoma") component
* Use of any investigational agent within 28 days prior to initiation of treatment
* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix within the last 5 years unless in complete remission since at least 3 years
* Dependency on red blood cell and/or platelet transfusions
* HBsAg positivity
* Evidence of central nervous system involvement
* A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
* Severe peripheral polyneuropathy
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months and/or long QT-syndrome
* HIV seropositivity
* Presence of active opportunistic infections
* Pregnancy or lactation
* Uncontrolled diabetes mellitus
* Pre-existing thromboembolic conditions at study entry
* Known hypersensitivity to thalidomide or lenalidomide or macrolide antibiotics
* Presence of any contraindication reported on the Summary of Product Characteristics (SmPC) of Clarithromycin
* Hypersensitivity to any active principle and/or any excipient according to the contraindications reported in the SmPC of clarithromycin and in the Investigator's Brochure (IB) of lenalidomide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Tumor response assessment | During the active treatment period after the 3rd cycles of both drugs administration
  The primary outcome measure is tumour response assessed according to the Revised Response Criteria for Malignant Lymphoma, either clinically (including appropriate imaging procedures) or endoscopically and histologically (in patients affected by gastric lymphoma, according to the GELA scoring system).

SECONDARY OUTCOMES:
Adverse Events assessments | During the active treatment period
  1. Treatment-emergent adverse events (AEs) incidence, severity and relationship to study treatment.
  2. Time from first IMP administration to assessment of disease progression or death due to any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Zucca, Prof, Study Director — International Extranodal Lymphoma Study Group
Locations (10):
- Medical University of Vienna, Vienna, Austria
- Italy (6):
  - A.O. Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Papardo, Messina
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Ospedale di Circolo e Fondazione Macchi di Varese, Varese
  - Azienda Sanitaria ULSS 6 - Ospedale S.Bortolo, Vicenza
- Spain (3):
  - Instituto de Enfermedades Hematológicas y Oncológicas, Barcelona, Barcellona
  - Institut Català D'Oncologia Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario, Salamanca

REFERENCES:
- [Derived] Pirosa MC, Sassone M, Kiesewetter B, Guillermo AL, Devizzi L, Domenech ED, Tucci A, Mannina D, Merli M, Salar A, Visco C, Esposito F, Bonomini L, Zucca E, Ferreri AJM, Raderer M. IELSG40/CLEO phase II trial of clarithromycin and lenalidomide in relapsed/refractory extranodal marginal zone lymphoma. Haematologica. 2023 Jun 1;108(6):1671-1675. doi: 10.3324/haematol.2022.281963. No abstract available. PMID 36546422